CLINICAL TRIAL: NCT05673837
Title: the Type ONe dIabetic Bone Collaboration Study
Acronym: TONICS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Odense University Hospital (Other)
Collaborators: Aalborg University Hospital (Other); Steno Diabetes Center Nordjylland (Other); Esbjerg Hospital - University Hospital of Southern Denmark (Other); Aarhus University Hospital (Other); Steno Diabetes Center Odense (Other); Molecular endocrinology department (KMEB) (Unknown)
Responsible Party: Principal Investigator, Inge Agnete Gerlach Brandt, Medical Doctor, PhD Student, Odense University Hospital
Other Study IDs: S-20200192
Record Dates: First submitted 2022-10-13; First posted 2023-01-06 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Osteoporosis Secondary; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Bone samples (from subgroup of 24+12 individuals), bone marrow aspirates(from subgroup of 24+12 individuals), blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Type 1 Diabetes: 111 persons with Type 1 Diabetes since childhood
- Controls: 37 persons without diabetes

SUMMARY:
In this cross-sectional clinical study, we will examine the bones of 111 Type 1 Diabetes (T1D) patients and 37 age-matched healthy controls with the aim of describing a T1D Bone Phenotype. The main Objectives of the study is a) to determine if the material properties of the bones are affected in diabetic bone disease and b) to determine if the mitochondrial function in osteoclasts and osteoblasts is impaired in T1D. Secondary end points are c) to establishment of the T1D bone phenotype and d) to investigate if mitochondrial dysfunction in T1D bone cells correlates to changes in gene expression, gene activity, bone remodelling, bone density, microarchitecture, geometry and material properties. Furthermore, in terms of contributing to knowledge on etiology and pathology of type one diabetic bone disease, we will study the predictory value of muscle mass in T1D patients and controls, as well as other characteristics such as heart rate variability (HRV) and AGE content. Furthermore, we will study the epidemiology of osteoporosis and fractures in Danish T1D patients.

To assess the material properties of the bones, we will measure the bone mass density (BMD), use High Resolution peripheral Quantitative Computed Tomography (HRpQCT) for assessment of the microarchitecture and finite element analysis of bone strength, and by microindentation, we will obtain direct measures of the strength of the cortical bone of the tibia. Further we will measure bone turnover markers and circulating microRNA and in a subgroup of participants (24 T1D, 12 controls) bone samples will be retrieved for examination of bone histomorphometry (structural and static parameters) and cell samples from blood and bone marrow will be used for in vitro experiments focused on cell differentiation mitochondrial function, as hyperglycemia may affect mitochondrial function. Finally measures of some possible predictors of bone fragility in subjects with T1D are examined (sarcopenia, skin advanced glycation end products (AGE) content, autonomic neuropathy)

DETAILED DESCRIPTION:
Methods The project consists of a cross-sectional case-control study bone histology, density and strength in adult T1D patients and in vitro studies of bone cell metabolism, including mitochondrial function in T1D.

Participants 111 male and female patients aged 18-80 years with early onset T1D (diagnosed before age of 18) and 37 healthy age-, sex- and BMI-matched control subjects. Of those 24 cases and 12 controls are needed for studies on bone biopsies and bone marrow aspirates.

Investigations Clinical data from digital medical records, survey and interview: c-peptide levels, medical history including information on diabetes-related complications, fracture history and concomitant medication.

Blood samples: hemoglobin A1c, ionized calcium (Ca2+), parathyroid hormone (PTH), 25-hydroxycholecalciferol, Hemoglobulin, Leucocytes, platelets, creatinin, estimated glomerular filtration rate (eGFR), Alkaline phosphatase, Alanine transaminase, albumin, international normalized prothrombin ratio (INR). And possibly c-peptide and T1D-related antibodies on T1D subjects, may these results not be found in the medical records. Fasting serum levels of biochemical markers of bone resorption, bone formation and inhibition of bone formation: Cross-linked C-telopeptide of type I collagen (CTX) Procollagen-1 N-terminal peptide (P1NP), Sclerostin, fasting levels of circulating miRNAs reported to be associated with bone turnover will be measured using quantitative PCR (qPCR) by use of a LightCycler 480 instrument (will be sent to measurement in Vienna (Dr M Hackl, TamiRNA, Vienna, Austria)).

For the participants that have accepted to have bone biopsy and marrow aspirate performed, we will measure Hemoglobulin, platelets, INR, activated partial thromboplastin time (APTT) 5 days prior to the biopsy. From these subjects, we will also obtain fullblood for: In vivo investigations on monocytes (osteoclastogenesis) and Resorption assays.

Dual-energy X-ray Absorptiometry (DXA) scan will provide BMD at the hip and spine as well as Trabecular Bone Score (TBS) and whole-body scan for a measure of muscle mass HR-pQCT at the distal radius and tibia, we will obtain: Bone geometry, Volumetric BMD, Bone microarchitecture, Bone strength.

by microindentation using OsteoProbe®, we will measure the material strength index (BMSi), a measure of the bone hardness and stiffness.

Bone biopsy: following bone labelling with oral tetracycline, an 8 mm trans iliac bone biopsy will be performed. Bone specimens will be plastic embedded and used for

* Bone histomorphometry (structural, static and dynamic parameters)
* Micro Finite Element Analysis (strength analysis)
* Ultra-high resolution measurements on osteocytes (number, density and connections)
* Immunohistochemistry and imaging for coupling factors and gene expression. Cryosectioned bone tissue will be used to perform spatial transcriptomics to assess the gene activity in bone-specific loci.

A Bone marrow aspirate 10-15 ml will be secured and used to study bone cells:

* Flowcytometric methods on in vitro studies on mesenchymal stem cells (MSCs) from bone marrow aspirates: expression, differentiation and proliferation to osteoblasts(OBs) and adipocytes.
* Monocytes from peripheral blood will be used to study osteoclastogenesis and bone resorption activity
* In vitro studies and proteomics of bone cell communication in co-cultures of OBs and osteoclast (OCs).
* Single cell RNA sequencing will be performed to demonstrate gene signatures of MSCs, OBs and OCs in T1D patients and controls.
* Determination of the metabolic profile (using the Seahorse Xfe96 Analyzer) and measurement of glucose uptake of MSCs, OBs and OCs in T1D patients and controls
* Imaging of mitochondrial morphology using MitoTracker.
* In situ hybridization and immunohistochemistry Outcome

Differences between early onset T1D patients and healthy age-matched controls in following parameters and the relationship between these parameters in T1D patients:

* BONE PHENOTYPE: Bone density, geometry, architecture, histomorphometry, ultra-high resolution measurements on osteocytes and finite element analysis (FEA) - calculated strength obtained from DXA scans, HRpQCT scans and from bone biopsies in a subgroup of the subjects and Bone hardness (Bone Score), measured by microindentation.
* BONE METABOLISM: Levels of skinAGEs and levels of biochemical bone turnover markers and circulating miRNA's known to be related to bone turnover, dynamic measures from bone histomorphometry. Immunohistochemistry and -imaging on bone biopsies.

In vitro analyses and other investigations on cells will produce outcomes on bone cell differentiation, proliferation and intercellular communication and coupling, bone cell gene signatures and metabolic profiles.

• PREDICTION VALUES of heart rate variability (Can assessment with Vagus(TM), skin autofluorescence (by AGE Reader from Diagnoptics) and muscle mass (by DXA whole-body scan) and - strength (by hand grip strength measured by dynamometer) Data will be summarized using odds ratios, trend analysis and regression analysis, adjusting for potential confounders. Students t-test and Chi square tests will be applied for test of group comparison. Statistical analyses will be conducted in Excel® and STATA®.

Power Calculation The total number of individuals that will be recruited is based on a previous study of bone strength in T2D patients (same method) showing bone material strength index (BMSi) of 78,2 (SD 7,5) in controls and 74,6 (SD 7,6) in T2D patients. With 111 T1D patients and 37 controls, the power of the study will be 80% to demonstrate a difference in bone strength of 4.

The number of participants needed for the studies on cell metabolism is based on an expected between-group difference in basal respiration of 25% when using the Seahorse extracellular flux analyser. (Difference of 25% is similar to that observed in another cell type in T1D and non-T1D patients in an on-going study at Aarhus University).

source data will be available on the scanners and as for other examinations, screenshots/photographs of result windows are saved in the encoded database, where the results are also typed in by hand.

Local monitoring will be carried out. Standard Operating Procedures for examinations are followed by involved clinicians and investigators.

ELIGIBILITY:
Inclusion Criteria:

* T1D subjects: Clinical diagnosis of T1D <18 years of age, C-peptide <200 pmol L-1 at any time point.
* Controls: HbA1c <44 mmol mol-1

Exclusion Criteria:

* BMI < 18.5 kg/m2
* Primary hyperparathyroidism and other calcium metabolic conditions
* Paget's disease and other metabolic bone diseases
* Vitamin D <25 nM (re-test after vitamin D replacement acceptable)
* Known disorders affecting bone metabolism, e.g. uncontrolled thyrotoxicosis, chronic kidney disease (eGFR <30 ml min-1), liver dysfunction (alkaline phosphatase higher than twice the upper limit), celiac disease not controlled by diet, known hypogonadism, severe chronic obstructive pulmonary disease, hypopituitarism and Cushing's disease
* Antiresorptive or bone metabolic drugs for the last 12 months
* Use of anabolic steroids in the last 12 months
* History of pancreatitis
* Allergy to the medicines used
* Inability to give informed consent
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Type 1 Diabetic subjects recruited from out-patient clinics and internet pages such as Facebook.
  Controls from community i.e. through advertisement on internet sites such as Facebook
Sampling Method: Non-Probability Sample
Enrollment: 148 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Mitochondrial function: oxygen consumption rate (OCR) | baseline
  using the Seahorse Xfe96 Analyzer and measurement of glucose uptake of MSCs, OBs and OCs
measurement of glucose uptake of MSCs, OBs and OCs | baseline
  using a bioluminescent assay (Glucose-Uptake Glo, Promega)
cell lactate production | baseline
  using the Seahorse Xfe96 Analyzer and measurement of glucose uptake of MSCs, OBs and OCs
Bone Material Strength index (BMSi) | baseline
  measure of microindentation on tibia by OsteoProbe(TM),. Measure given as index: BMSi. The strength of the bone is higher with higher BMSi measures which measures from approx. 40 to 90 (no unit)
Bone mineral density by DXA | baseline
  DXA scan of hip and spine
Spine trabecular bone score (TBS) | baseline
  estimated by software of DXA on spine using Hologic Horizon A. Approx. 1000 to 1600 with higher quality of the network with higher values of TBS
Cortical thickness(Ct.Th) | baseline
  measured By High Resolution periphery Quantitative Computed Tomography(HRpQCT)
Failure load | baseline
  measured Finite Element Analysis by High Resolution periphery Quantitative Computed Tomography(HRpQCT)
volumetric Bone material density (vBMD) | baseline
  measured By High Resolution periphery Quantitative Computed Tomography(HRpQCT)

SECONDARY OUTCOMES:
microRNA and gene network analyses | baseline
  Gene expression and activity in cell samples from blood and bone marrow by established methods and including analyses of microRNA and gene network analyses
microarchitecture | baseline
  By ultramicroscopy of histologic bone samples, the microarchitecture can be analyzed and compared in the case and control groups
Mineralizing surface (MS/BS, %) | baseline
  By analyses of bone histomorphometry in the case and control groups as a measure of the bone remodelling in T1D bones
Mineral apposition rate (MAR micrometer/day) | baseline
  By analyses of bone histomorphometry in the case and control groups as a measure of the bone remodelling in T1D bones
Bone formation rate (BFR/BS) | baseline
  By analyses of bone histomorphometry in the case and control groups as a measure of the bone remodelling in T1D bones
bone turnover markers | baseline
  By analyses of bone bone turnover markers P1NP, CTX and sclerostin and comparison of the the case and control groups we will analyse the bone remodelling in T1D bones
Tb bone volume fraction (BV/TV) | baseline
  measured By High Resolution periphery Quantitative Computed Tomography(HRpQCT)
Trabecular thickness (Tb.Th) | baseline
  measured By High Resolution periphery Quantitative Computed Tomography(HRpQCT)
Cortical porosity(Ct.Po) | baseline
  measured By High Resolution periphery Quantitative Computed Tomography(HRpQCT)
skin autofluorescence (SAF) | baseline
  measured by AGE Reader(R) as a surrogate marker for bone AGE content. measures from appr. 0.5 to 4.5 (no unit). The higher the value the greater the tissue accumulation of fluorescent advanced glycation end products
Handgrip Strength | baseline
  Handgrip Strength in kg measured with hydraulic HandGrip Dynamometer as one of two measures of sarcopenia
Lean mass | baseline
  Estimated lean mass from DXA wholebody scan as one of two measures of sarcopenia
Cardiologic Autonomic Neuropathy measure (CAN) | baseline
  by Vagus (TM) as a measure of autonomic neuropathy which returns CAN score of 0 or zero in each of three measurements (rise up, deep breathing and valsalva manoeuvre), calculating a total CAN score of 0 to 3 where 0 is no CAN, 1 is borderline CAN and 2 is a positive CAN screening.
Trabecular spacing (Tb.Sp) | baseline
  measured By High Resolution periphery Quantitative Computed Tomography(HRpQCT)
Trabecular area | baseline
  measured By High Resolution periphery Quantitative Computed Tomography(HRpQCT)

OTHER OUTCOMES:
Cortical area | baseline
  measured By High Resolution periphery Quantitative Computed Tomography(HRpQCT)
Endosteal perimeter | baseline
  measured By High Resolution periphery Quantitative Computed Tomography(HRpQCT)
Periosteal perimeter | baseline
  measured By High Resolution periphery Quantitative Computed Tomography(HRpQCT)
Bone Stiffness | baseline
  measured Finite Element Analysis by High Resolution periphery Quantitative Computed Tomography(HRpQCT)
Trabecular Thickness (Tb.Th) | baseline
  measured By High Resolution periphery Quantitative Computed Tomography(HRpQCT)
Trabecular number (Tb.N) | baseline
  measured By High Resolution periphery Quantitative Computed Tomography(HRpQCT)
Other structural and remodelling measures from bone histomorphometry | baseline
  Osteoid surface (OS/BS, %), Osteoblast surface (Ob.S/BS) and Eroded surface (ES/BS, %)

CONTACTS AND LOCATIONS:
Overall Officials: Morten F Nielsen, MD PhD Prof., Principal Investigator — Odense University Hospital
Locations (1):
- Steno Diabetes Center Nordjylland, Aalborg, Denmark